CLINICAL TRIAL: NCT03198923
Title: A Phase 1/2 Safety and Efficacy Study of Natural Killer and Natural Killer T Cell Immunotherapy in Patients With Non Small Cell Lung Cancer
Brief Title: Clinical Efficacy and Safety of NK and NKT Cells Infusion in Patients With Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenxiang Wang (Other)
Collaborators: Shanghai Houchao Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Wenxiang Wang, Professor, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKNKTLC001
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- natural killer and natural killer T cell (Experimental): The eligible patients are infused with ten doses of (2-2.5)x10^9 NK and NKT cells in one course of treatment.
  Interventions: Biological: natural killer and natural killer T cell

INTERVENTIONS:
Biological: natural killer and natural killer T cell — The eligible patients are infused with 10 doses of (2-2.5)x10^9 NK and NKT cells in one course of treatment.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of natural killer (NK) cell and natural killer T (NKT) cell-based immunotherapy in subjects with non small cell lung cancer.

DETAILED DESCRIPTION:
With the development of oncology and immunology in recent years, immunotherapy represents a novel path to obtain a durable and long-lasting response in cancer patients. NK and NKT cells are expanded conventionally from peripheral blood mononuclear cells by addition of a variety of cytokines in vitro culture. Our previous studies demonstrated that the expansion of NK and NKT cells in a clinical usage scale from peripheral blood mononuclear cells is feasible. Those expanded NK and NKT cells exhibit antitumor effect in vitro and in vivo against a variety of tumor cells. The current study proposes a 3-course treatment of doses administered at one week intervals with monitoring at each administration plus 4 weeks after the last dose. The total study time (apheresis through last follow-up) is estimated at 3 year.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years, Male or Female
* Histological or cytologically diagnosis of non-small cell lung cancer
* Recurrent or metastatic after surgical treatment
* The pathology must be an assessable disease, signal lesion not exceeding 3 cm in diameter (measurable by CT scan or MRI)，number of Lymph node metastasis is less than 5
* Refractory to standard treatments (e.g., chemotherapy, radiation, etc.)
* No chemotherapy and radiation therapy to be planned recently
* Patients must have a Karnofsky performance status greater than or equal to 70%
* Life expectancy greater than 3 months
* Able and willing to give witnessed, written informed consent form prior to receiving any study related procedure
* Agree that progress of the disease must be radiographically measurable by computerized tomography (CT) scanning technique or magnetic resonance imaging (MRI) (per RECIST1.1 criteria)
* Agrees to participate in long-term follow-up for up to 3 years, if received NK and NKT infusion
* Laboratory values within the following ranges prior to receiving treatment of study agent: Peripheral blood cells >3×10^9 /L; Number of lymphocytes >1.0×10^9 /L; Lymphocyte ratio >18%; INR<1.5.

Exclusion Criteria:

* Patients with no surgical treatment
* Patients within concurrent chemotherapy or radiation
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Negative HIV antigen and antibody, Hepatitis B surface antigen and Hepatitis C PCR within 21 days prior to enrollment
* History of immunodeficiency disease or autoimmune disease
* Patients with chronic disease which is undergoing immune reagents or hormone therapy
* Serious infections requiring antibiotics, bleeding disorders
* Previous bone marrow or stem cell transplant, or organ allograft
* Concurrent other medical condition that would prevent the patient from undergoing protocol-based therapy
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent
* Pregnant or breast-feeding patients
* Lack of availability of a patient for immunological and clinical follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events following infusion of NK and NKT cells | 30 days post-infusion
Overall Survival (OS) | Approximately 3 years

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Approximately 1 years
Objective Response Rate (ORR) | up to 24 weeks
  confirmed by CT or MRI, or confirmed by biopsy
Tumor Marker | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenxiang Wang, PhD, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No